CLINICAL TRIAL: NCT02913209
Title: Quantitative Fatigue and Muscle Performance in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Harris-Love, Assoc. Director of the CRC Human Performance Research Unit, Washington D.C. Veterans Affairs Medical Center
Other Study IDs: MRIB 01772
Record Dates: First submitted 2016-08-02; First posted 2016-09-23 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple Sclerosis Fatigue (MSF) Cohort: Participants will complete study assessments over 4 visits to the DC VAMC. Disease severity will be assessed by the EDSS, and a cognitive battery will be completed. Peak torque assessment for the knee flexors and extensors will be performed on an isokinetic dynamometer (Biodex System 4). Muscle morphology measures of the rectus femoris will be obtained using diagnostic musculoskeletal ultrasound. The sonographic measures will include muscle thickness and echogenicity. Isokinetic and isoinertial mode fatigue measures for the knee extensors will be assessed on separate visits (at least 48 hours apart). Performance-based measures of function will include an assessment of patient mobility and the 25-foot walk test. Muscle power will be estimated by the timed sit to stand test. Subjective measures of fatigue and quality of life include the MSQoL, MFIS, and Neurology Quality of Life Adult Fatigue Bank (AFB).

SUMMARY:
Fatigue is consistently rated as the top symptomatic complaint for individuals with multiple sclerosis (MS). Currently, the MS Fatigue Impact Scale (MFIS), a subsection of the Multiple Sclerosis Quality of Life (MSQoL), is the clinical standard used by neurologists for monitoring and tracking fatigue in individuals with MS. However, fatigue is multidimensional phenomenon and subjective measures have had poor or limited relationships with functional status. While previous study has focused on contributing factors to fatigue such as sleep disorders and diminished cortical excitability, this line of inquiry has neglected the role of muscle structure and function on fatigue in every day functional tasks. An alternative approach is to assess quantitative fatigue using anaerobic testing methods. However, more knowledge is needed to understand the role that quantitative fatigue plays in self-reported fatigue measures and function of daily activities. Our purpose is to determine the association between quantitative fatigue tests with performance-based measures of mobility and self-reported health-related quality of life. Our secondary goal is to understand how the intrinsic properties of muscle tissue influence muscle performance in Veterans with MS.

DETAILED DESCRIPTION:
Participants will complete study assessments at the DC VAMC. Disease severity will be assessed by medical staff completing the EDSS. Peak torque assessment for the knee flexors and extensors will be performed on an isokinetic dynamometer (Biodex System 4). Muscle morphology measures of the rectus femoris will be obtained using diagnostic musculoskeletal B-mode ultrasound (Phillips EPIQ 7 180 Plus) with a 10 Mhz linear transducer. The sonographic measures will include muscle thickness and echogenicity. The mode of exercise testing and the type of muscle action will influence the assessment of fatigue. Therefore, isokinetic fatigue measures for the knee extensors will be assessed on separate visits (at least 48 hours apart). Performance-based measures of function will include an assessment of patient mobility and the 25-foot walk test. Muscle power will be estimated by the timed sit to stand test. Subjective measures of fatigue and quality of life include the MSQoL, MFIS, and Neurology Quality of Life Adult Fatigue Bank (AFB).

ELIGIBILITY:
Inclusion Criteria:

* A male or female Veteran participant must have a medical diagnosis of multiple sclerosis
* Veteran will be between the ages of 20 and 85 years old

Exclusion Criteria:

* Veterans with an EDSS score > 7.0
* Veterans with any cardiac condition that may cause sudden decompensation during exertional fatigue testing (e.g., severe congestive heart failure and uncontrolled hypertension)
* Veterans found to have severe depression (BDI score >28)
* Veterans with lower extremity amputation
* Steroid Infusion less than 2 weeks prior to enrollment
* Veterans with a lower extremity joint replacement
* Veterans that exhibit severe cognitive impairment
* Defined as loss of orientation to person, place and/or time and an inability to follow three step commands.
* Veterans that are unable to perform a stand pivot transfer with minimal assist

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women between the ages of 20 and 85 years (n=30) with a history of multiple sclerosis (Expanded Disability Status Scale, EDSS < 7.0) will be consecutively recruited from the DC VAMC Neurology Service and Multiple Sclerosis Center of Excellence.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2018-10 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue Index | Day 1
  Initial visit
Maximal Volitional Contraction | Day 1
  Initial visit

SECONDARY OUTCOMES:
The Adult Myopathy Assessment Tool | Day 1
  Initial visit
25 foot walk Test | Day 1
  Initial visit
Chair Stand Test | Day 1
  Initial visit
Modified Fatigue Impact Scale | Day 1
  Initial visit
Multiple Sclerosis Quality of Life | Day 1
  Initial visit
Adult Fatigue Bank | Day 1
  Initial visit
Ultrasound caliper measure of rectus femoris thickness | Day 1
  Initial visit
Ultrasound image post-processing of rectus femoris grayscale | Day 1
  Initial visit

OTHER OUTCOMES:
Kurtzke Expanded Disability Status Scale | Day 1
  Initial visit

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, DSc, Principal Investigator — Washington DC VA Medical Center

REFERENCES:
- [Background] Seamon BA, Harris-Love MO. Clinical Assessment of Fatigability in Multiple Sclerosis: A Shift from Perception to Performance. Front Neurol. 2016 Nov 7;7:194. doi: 10.3389/fneur.2016.00194. eCollection 2016. No abstract available. PMID 27872608